CLINICAL TRIAL: NCT06522139
Title: Clinical Outcome After Episealer Talus Implant in Treatment of Osteochondral Lesion of the Talus
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stefano Zaffagnini (Other)
Responsible Party: Sponsor-Investigator, Stefano Zaffagnini, Principal Investigator, Istituto Ortopedico Rizzoli
Organization: Istituto Ortopedico Rizzoli (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Epi-Talus
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Osteochondral Defect
Keywords: Talus Osteotomy; Osteochondral lesion; foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sperimental (Experimental): Implantation of Episealer Talus Implant
  Interventions: Procedure: Implantation of Episealer Talus Implant

INTERVENTIONS:
Procedure: Implantation of Episealer Talus Implant — Subjects will be on study for up to 60 months after their talus implant surgery. Treatment: Implantation of Episealer Talus Implant Follow-up: 60 months The total duration of the study is expected to be 75 months. 12 months for subject recruitment, 60 for final subject follow-up and 3 for data analysis and production of the final report.

SUMMARY:
Autologous Chondrocyte Implantation (ACI) is an appealing technique whereby cartilage is harvested from the joint in a first operation. This biopsy is processed, individual cells are freed and cultivated and, in a second procedure, injected into the defect that has been covered by a periosteal graft). A second generation includes a matrix (MACI) into which the cells are injected/cultivated. Recently, collagen membranes are used to cover the cells or cover a micro-fractured defect. Good results have been reported although return to previous sports remains a challenge . Long term results are lacking. More important is the fact that these treatments are directed towards restoring the articular cartilage whereas the patient's symptoms are generated by the bone and not the cartilage.

Treatment of an OCD with a small metallic implant has been tested in recent years. Results have been promising by some reports, while a high revision rates was reported by others. A recent 2-8 years follow-up study revealed a survival rate of 95 %

ELIGIBILITY:
Inclusion Criteria:

* Osteochondral lesion (both primary and secondary lesions) ⌀ 10-15 mm on the medial or lateral talar dome
* age between 18 and 65 years
* BMI < 35
* patients who have given their willingness to reach the Institute for checkups.
* patients previously treated with conservative therapies, which proved unsuccessful

Exclusion Criteria:

* non-focal defect
* on-going infection in the ankle joint
* inflammatory arthritis or radiographic osteoarthritis in the ankle joint (=no joint space narrowing) Osteophytes without joint space narrowing (=Gr1 (van Dijk classification)) is not a contra indication.
* sensitivity to cobalt-chrome alloys and titanium materials
* inadequate bone stock where the Episealer is to be inserted
* existing prosthesis in the area of treatment or opposing surface
* osteochondral lesion on opposing tibial surface
* pain of unknown etiology
* demineralised bone
* instability. Instability is defined as recurrent giving way with or without laxity
* severe malalignment in the ankle joint >5 degrees malalignment as compared to the contralateral ankle joint, as measured on the standing X-Ray
* Ipsilateral symptomatic foot, knee or hip disease which affects the mobility of the patient
* other diseases or medication that may affect the bone anchoring of the Episealer
* uncooperative patient that is not willing to follow instructions
* muscular insufficiency
* vascular insufficiency
* medical, hormonal, hematological, immunological or metabolic illnesses
* Smoking
* Pregnancy
* Diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
FOOT AND ANKLE OUTCOME SCORE -symptoms | after 12 months from the intervention
  The FAOS (Foot and Ankle outcome score) is a 42-item questionnaire, 7 items for symptoms
Implant survival | after 5 years
  Implant survival rate at 60 months follow-up
FOOT AND ANKLE OUTCOME SCORE - pain | after 12 months from the intervention
  The FAOS (Foot and Ankle outcome score) is a 42-item questionnaire, 9 for pain
FOOT AND ANKLE OUTCOME SCORE -symptoms | after 24 months from the intervention
  The FAOS (Foot and Ankle outcome score) is a 42-item questionnaire, 7 items for symptoms
FOOT AND ANKLE OUTCOME SCORE - Pain | after 24 months from the intervention
  The FAOS (Foot and Ankle outcome score) is a 42-item questionnaire, 9 for pain

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy